CLINICAL TRIAL: NCT02499796
Title: Short-term Effects of Humidification Devices on Respiratory Pattern and Work of Breathing During Invasive Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Annia Schreiber, MD, Fondazione Salvatore Maugeri
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 981
Record Dates: First submitted 2015-07-08; First posted 2015-07-16 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Chronic Respiratory Failure
Keywords: Invasive mechanical ventilation; Humidifying devices; Respiratory mechanics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Every patient receives 20 minutes of invasive mechanical ventilation with each of the three humidification systems in random sequence:
  * Heated and moisture exchanger (HME)
  * Heated humidifier (HH)
  * Hygrovent Gold
  Interventions: Device: Hygrovent Gold; Device: Heated and moisture exchanger (HME); Device: Heated humidifier (HH)

INTERVENTIONS:
Device: Hygrovent Gold
Device: Heated and moisture exchanger (HME)
Device: Heated humidifier (HH)

SUMMARY:
This study compares the short-term effects of a new humidification system (Hygrovent Gold) and two other humidification devices (heated and moisture exchanger and heated humidifier) on respiratory pattern and work of breathing, during invasive ventilation.

DETAILED DESCRIPTION:
Three humidifying devices are commonly and indifferently used during mechanical ventilation, but their impact on respiratory mechanics and, eventually, mechanical ventilation efficacy, particularly in patients highly dependent from mechanical ventilation, are not superimposable.

It has already been described that heated and moisture exchangers (HME), increasing dead space, can negatively affect ventilatory function and gas exchange, in comparison to heated humidifiers (HH).

The Hygrovent Gold, mainly because of its position between the tracheostomy and the Y-piece of the ventilatory circuit and its structure, may lead to analogous or even worse effects, determining and increase in inspiratory resistances and dead space and consequently an increase in the work of breathing.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hypercapnic respiratory failure (PaCO2 of 45 mmHg or more)
* Long-term mechanical ventilation via tracheostomy
* Clinical stability

Exclusion Criteria:

* Non collaborative subjects
* Acute respiratory failure
* Haemodynamic instability
* Encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in muscle pressure-time product (PTPoes) | Baseline and 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ceriana, MD, Study Chair — Fondazione Salvatore Maugeri
Locations (1):
- Fondazione Salvatore Maugeri, Pavia, Italy

REFERENCES:
- [Background] Lellouche F, Maggiore SM, Deye N, Taille S, Pigeot J, Harf A, Brochard L. Effect of the humidification device on the work of breathing during noninvasive ventilation. Intensive Care Med. 2002 Nov;28(11):1582-9. doi: 10.1007/s00134-002-1518-9. Epub 2002 Oct 10. PMID 12415444
- [Background] Jaber S, Chanques G, Matecki S, Ramonatxo M, Souche B, Perrigault PF, Eledjam JJ. Comparison of the effects of heat and moisture exchangers and heated humidifiers on ventilation and gas exchange during non-invasive ventilation. Intensive Care Med. 2002 Nov;28(11):1590-4. doi: 10.1007/s00134-002-1441-0. Epub 2002 Sep 6. PMID 12415445
- [Derived] Schreiber AF, Ceriana P, Ambrosino N, Piran M, Malovini A, Carlucci A. Short-Term Effects of an Active Heat-and-Moisture Exchanger During Invasive Ventilation. Respir Care. 2019 Oct;64(10):1215-1221. doi: 10.4187/respcare.06799. Epub 2019 Jul 3. PMID 31270176